CLINICAL TRIAL: NCT05891132
Title: Comparison Between the Effects of Lidocaine Prilocaine Cream and Lidocaine Injection on Reduction of Perineal Pain During Episiotomy and Perineum Repair in Vaginal Delivery: Randomized Control Trial
Brief Title: Comparison Between Lidocaine Prilocaine Cream and Lidocaine Injection on Pain Control During Episiotomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed ElHarty, lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-12-2023
Record Dates: First submitted 2023-05-26; First posted 2023-06-06 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Episiotomy Wound
Keywords: Episiotomy; Anesthesia during labor; Injectable anesthetic; Topical anesthetic; Postpartum pain; Postpartum infection; Dyspareunia
MeSH Terms: conditions — Dyspareunia | interventions — Injections; Anesthetics; Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Intervention Model Description: Group I comprised 30 women who will receive 10 ml of lidocaine 2% for perineal infiltration at the time of crowning while 30 women.
  Group II will have lidocaine prilocaine cream 15gm application on the perineum at 8 cm of cervical dilatation and then additional dose every 1 hour until delivery is achieved, then another dose of the cream will be applied before repairing the episiotomy and finally daily 3 doses every 8 hours at the site of episiotomy for the first week post-partum.
Who Masked: Participant
Masking Description: This will be a randomized controlled trial, randomization will be achieved by the following: the allocation treatment will be written on cards that will be sealed in sequentially numbered envelopes. The envelopes will be opened at the time of allocation after the enrolled participants will complete all baseline assessments. Group I comprised 30 women who will receive 10 ml of lidocaine 2% for perineal infiltration at the time of crowning while 30 women of Group II will have lidocaine prilocaine cream 15gm application on the perineum at 8 cm of cervical dilatation and then an additional dose every 1 hour until delivery is achieved, then another dose of the cream will be applied before repairing the episiotomy and finally daily 3 doses every 8 hours at the site of episiotomy for the first week post-partum.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I comprised 30 women who will receive 10 ml of lidocaine 2% (Active Comparator): 10 ml of lidocaine 2% for perineal infiltration at the time of crowning
  Interventions: Drug: 10 ml of lidocaine 2%
- Group II will have lidocaine prilocaine cream 15gm application on the perineum (Active Comparator): lidocaine-prilocaine cream 15gm application on the perineum at 8 cm of cervical dilatation and then an additional dose every 1 hour until delivery is achieved, then another dose of the cream will be applied before repairing the episiotomy and finally daily 3 doses every 8 hours at the site of episiotomy for the first week post-partum
  Interventions: Drug: lidocaine prilocaine cream 15gm

INTERVENTIONS:
Drug: 10 ml of lidocaine 2% — 10 ml of lidocaine 2% for perineal infiltration at the time of crowning
  Other Names: Local ( injectable ) anesthetic
  Arms: Group I comprised 30 women who will receive 10 ml of lidocaine 2%
Drug: lidocaine prilocaine cream 15gm — Lidocaine prilocaine cream, an eutectic mixture, is composed of Lidocaine-25 mg, Prilocaine-25 mg, Arlactone 289 -19 mg, Carbopol-10 mg, Sodium hydroxide to make a pH of 9.6 mg and purified water to produce l gram.
  Other Names: EMLA cream
  Arms: Group II will have lidocaine prilocaine cream 15gm application on the perineum

SUMMARY:
The present study aims to compare the effects of lidocaine-prilocaine cream and lidocaine injection on the reduction of pain while doing and repairing episiotomy, controlling the pain in the post-partum period, and reduction the risk of infection in 6 weeks post partum and dyspareunia after 6 weeks post-partum.

DETAILED DESCRIPTION:
Population of study & disease condition:

The study will be conducted on 60 patients that will be admitted to the labor ward in the Department of Obstetrics & Gynecology of a tertiary care center of Cairo University from Jan/2023 to Jan/2024 on. Primigravida women with singleton live pregnancy with cephalic presentation in the first stage of labor will be included in the study after approval by the Institutional Ethical Committee and obtaining an informed consent. Those with known allergy to lignocaine, altered mental status, request for epidural analgesia and hepatic disorders will be excluded from the study. The enrolled women will be divided into two groups by simple randomization with a 1:1 allocation ratio.

The following will be done to all participants:

* Informed written consent: after discussing the nature of the study as well as the expected value, outcome, and possible adverse effects.
* Full medical history: including full obstetric history and current pregnancy history (entailing the 1st day of LMP).
* Thorough Clinical Examination: general (vital signs) and full obstetric examination.
* Obstetric ultrasonography: to confirm gestational age and the eligibility of the current pregnancy to participate in the study.

This will be a randomized controlled trial, randomization will be achieved by the following: the allocation treatment will be written on cards that will be sealed in sequentially numbered envelopes. The envelopes will be opened at the time of allocation after the enrolled participants will complete all baseline assessments. Group I comprised 30 women who will receive 10 ml of lidocaine 2% for perineal infiltration at the time of crowning while 30 women of Group II will have lidocaine prilocaine cream 15gm application on the perineum at 8 cm of cervical dilatation and then additional dose every 1 hour until delivery is achieved, then another dose of the cream will be applied before repairing the episiotomy and finally daily 3 doses every 8 hours at the site of episiotomy for the first week post-partum. Lidocaine prilocaine cream, an eutectic mixture, is composed of Lidocaine-25 mg, Prilocaine-25 mg, Arlactone 289 -19 mg, Carbopol-10 mg, Sodium hydroxide to make a pH of 9.6 mg and purified water to produce l gram.

Fifteen grams of this cream will be applied as a thick layer (about 2 g/ 10 cm2 area) to the intact surface of the perineum and will be covered with an occlusive dressing (Kumar et al., 2015).

In previous study done by Nirmala et al., 2013 The mean pain scores in the study were comparable for both groups, in our study we will increase the dose and the intervals of the applied cream and we will write down the results regarding pain score and side effects.

At the time of crowning, the occlusive dressing and any residue of the cream will be removed and episiotomy will be done. The request for additional anesthetic agent (10 ml of 2% lidocaine solution for both groups) will be honored and recorded for both groups. And if the patient require additional analgesia during episiotomy (VAS more than 3) we will give additional anesthetic agent (10 ml of 2% lidocaine solution. After the repair of episiotomy, each patient will be asked to grade the severity of pain during perineal repair on a Visual Analog Scale (VAS). The far left will be labeled 'No pain' and the far right will be labelled as 'worst pain possible'. The subject will be asked to make a vertical mark on this line reflecting the severity of the pain.

The patients are followed 6 weeks post-partum at the OPC or by telephone call to check the pain score by using CAST score (Very satisfied - satisfied - not satisfied - dissatisfied).

Post-operative analgesics will include Paracetamol mainly and adjuvant NSAIDs as mentioned in the step ladder pain management by the WHO.

If any further analgesia needed we will use Pethidine as a rescue analgesic as it is safe after delivery but we will prescribe anti emetic with pethidine as it will induce nausea and vomiting.

Pain score during episiotomy repair will be the primary outcome of the study. Secondary outcome measures will include pain score in the first six weeks post-partum, dyspareunia after 6 weeks post-partum ( return to sexual life ) and reduction of the rate of wound infection.

Study location:

Kasr Al Ainy - Causality department (Department 10).

what does research involve? Human participants

Type of consent of study participants:

Written consent

Confidentiality of data:

- All study-related information will be stored at the study site.

Type of the study:

- Randomized Control Trial (RCT)

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women candidate for VD ( ASA Ⅱ )
2. Primigravida
3. Pregnant more than 37 weeks (Term pregnancy).
4. Singleton fetus.
5. Cephalic presentation.
6. In first stage of labor.

Exclusion Criteria:

1. More than or equal 1 previous CS and VBAC.
2. Multiparous women.
3. Pregnant less than 37 weeks
4. Twin pregnancy.
5. Not in active labor
6. allergy to lignocaine
7. altered mental status
8. request for epidural analgesia
9. Hepatic impairment.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-07-19 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Effect of the Intervention on pain score during the repair of episiotomy | 1 year
  Efficacy of lidocaine-pridocaine cream in pain control for episiotomy incision and repair assessed by Visual Analogue Score VAS during episiotomy incision and repair where the minimum value is equal to zero which means no pain at all and the maximum value is equal to 10 and this means the worst pain ever.

SECONDARY OUTCOMES:
Effect of the Intervention on pain score during 6 weeks postpartum and dyspareunia after 6 weeks post partum | 1 year
  Pain score in the first week post-partum and 6 weeks post-partum also dysparunia after 6 weeks of delivery will be assessed by Customer Satisfaction Score or CSAT score, where the minimum value is very unsatisfied and associated with the highest degree of pain and the maximum value is very satisfied and this associated with the lowest degree of pain in 1 week and 6 weeks post patum
Effect of the Intervention on perineal infection during 6 weeks postpartum | 1 year
  Detection of the infection rates 6 weeks post-partum as this is the period of perpurium when puerperal sepsis may develops.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Alharty, MD, Study Director — Cairo U
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Not for IPD

REFERENCES:
- [Background] Dahlen HG, Homer CS, Cooke M, Upton AM, Nunn RA, Brodrick BS. 'Soothing the ring of fire': Australian women's and midwives' experiences of using perineal warm packs in the second stage of labour. Midwifery. 2009 Apr;25(2):e39-48. doi: 10.1016/j.midw.2007.08.002. Epub 2007 Nov 26. PMID 18031878
- [Background] East CE, Sherburn M, Nagle C, Said J, Forster D. Perineal pain following childbirth: prevalence, effects on postnatal recovery and analgesia usage. Midwifery. 2012 Feb;28(1):93-7. doi: 10.1016/j.midw.2010.11.009. Epub 2011 Jan 13. PMID 21236531
- [Background] El-Boghdadly K, Pawa A, Chin KJ. Local anesthetic systemic toxicity: current perspectives. Local Reg Anesth. 2018 Aug 8;11:35-44. doi: 10.2147/LRA.S154512. eCollection 2018. PMID 30122981
- [Background] Field T. Pregnancy and labor alternative therapy research. Altern Ther Health Med. 2008 Sep-Oct;14(5):28-34. PMID 18780582
- [Background] Simionescu R. [Stress reaction and anesthesia. The role of morphine agonists and antagonists]. Cah Anesthesiol. 1988 Jun-Jul;36(4):289-301. No abstract available. French. PMID 3048583
- [Background] Jorge LL, Feres CC, Teles VE. Topical preparations for pain relief: efficacy and patient adherence. J Pain Res. 2010 Dec 20;4:11-24. doi: 10.2147/JPR.S9492. PMID 21386951
- [Background] Kargar R, Aghazadeh-Nainie A, Khoddami-Vishteh HR. Comparison of the Effects of Lidocaine Prilocaine Cream (EMLA) and Lidocaine Injection on Reduction of Perineal Pain During Perineum Repair in Normal Vaginal Delivery. J Family Reprod Health. 2016 Mar;10(1):21-6. PMID 27385970
- [Background] Lullmann B, Leonhardt J, Metzelder M, Hoy L, Gerr H, Linderkamp C, Klein C, Grigull L. Pain reduction in children during port-a-cath catheter puncture using local anaesthesia with EMLA. Eur J Pediatr. 2010 Dec;169(12):1465-9. doi: 10.1007/s00431-010-1244-1. Epub 2010 Jul 10. PMID 20623233
- [Background] Sanders J, Peters TJ, Campbell R. Techniques to reduce perineal pain during spontaneous vaginal delivery and perineal suturing: a UK survey of midwifery practice. Midwifery. 2005 Jun;21(2):154-60. doi: 10.1016/j.midw.2004.12.003. Epub 2005 Mar 27. PMID 15878430
- [Background] Shahrahmani H, Kariman N, Jannesari S, Rafieian-Kopaei M, Mirzaei M, Ghalandari S, Shahrahmani N, Mardani G. The effect of green tea ointment on episiotomy pain and wound healing in primiparous women: A randomized, double-blind, placebo-controlled clinical trial. Phytother Res. 2018 Mar;32(3):522-530. doi: 10.1002/ptr.5999. Epub 2017 Dec 13. PMID 29235159
- [Background] Shavit I, Hadash A, Knaani-Levinz H, Shachor-Meyouhas Y, Kassis I. Lidocaine-based topical anesthetic with disinfectant (LidoDin) versus EMLA for venipuncture: a randomized controlled trial. Clin J Pain. 2009 Oct;25(8):711-4. doi: 10.1097/AJP.0b013e3181a689ec. PMID 19920722
- [Background] Greveling K, Prens EP, Liu L, van Doorn MBA. Non-invasive anaesthetic methods for dermatological laser procedures: a systematic review. J Eur Acad Dermatol Venereol. 2017 Jul;31(7):1096-1110. doi: 10.1111/jdv.14130. Epub 2017 Feb 8. PMID 28107576
- [Background] Walker SM. Neonatal pain. Paediatr Anaesth. 2014 Jan;24(1):39-48. doi: 10.1111/pan.12293. Epub 2013 Nov 13. PMID 24330444
- [Background] Zilbert A. Topical anesthesia for minor gynecological procedures: a review. Obstet Gynecol Surv. 2002 Mar;57(3):171-8. doi: 10.1097/00006254-200203000-00022. PMID 11889416
- See also: An investigation into the effect of alpha ointment (fundermol) on perineal pain relief following episiotomy in Nulliparous Women — https://jmrh.mums.ac.ir/article_7979.htmlhttp://jmrh.mums.ac.ir/article_9975.html
- See also: Comparative study of eutectic mixture of lignocaine-prilocaine (EMLA) cream and lignocaine infiltration for pain relief during episiotomy and its repair — http://articles.theindianpractitioner.com/index.php/tip/article/view/158
- See also: Who invented the episiotomy? On the history of the episiotomy — https://europepmc.org/article/med/8503239
- See also: Comparison between lidocaine-prilocaine cream (EMLA) and Mepivacaine infiltration for pain relief during perineal repair after childbirth: A randomized trial. American Journal of Obstetrics and Gynecology, 201(2). — https://doi.org/10.1016/j.ajog.2009.04.023
- See also: Kumar, M., Chawla, R., & Goyal, M. (2015). Topical anesthesia. Journal of Anaesthesiology Clinical Pharmacology, 31(4), 450 — https://doi.org/10.4103/0970-9185.169049
- See also: Macarthur, A. J. & Macarthur, C. Incidence, severity, and determinants of perineal pain after vaginal delivery: A prospective cohort study. American Journal of Obstetrics and Gynecology 191, 1199-1204 (2004). — https://doi.org/10.1016/j.ajog.2004.02.064
- See also: Nirmala D, Ritu NA: ndalTopical lidocaine- prilocaine cream versus lignocaine infiltration for episiotomy repair: A randomized clinical trial. (2013). Journal of Clinical Research & Governance. — https://scholar.archive.org/work/fatlevhx3jbm7j6qoe63wutrey/access/wayback/http://index.sciencepub.se/ojs/index.php/JCRG/article/download/59/27